CLINICAL TRIAL: NCT00077025
Title: Phase II Multicenter, Double-Blind, Randomized Trial Comparing Anastrozole (ZD1033, Arimidex™)-Placebo to the Combination Anastrozole-ZD1839 (Gefitinib, IRESSA™) in Postmenopausal Patients With Estrogen Receptor (ER) and/or Progesterone Receptor (PgR) Metastatic Breast Cancer
Brief Title: Comparing Anastrozole-Placebo to the Combination Anastrozole-ZD1839 in Postmenopausal Patients With Estrogen Receptor and/or Progesterone Receptor Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1839US/0713
Record Dates: First submitted 2004-02-09; First posted 2004-02-11 (Estimated); Last update posted 2014-07-16 (Estimated); Status verified 2014-07

CONDITIONS: Breast Cancer
Keywords: metastatic breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Gefitinib; Anastrozole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Anastrozole-placebo (Active Comparator): Anastrozole (ZD1033, Arimidex)-Placebo
  Interventions: Drug: Anastrozole
- Anastrozole-ZD1839 (Active Comparator): Anastrozole (ZD1033, Arimidex)-ZD1839 (gefitinib, IRESSA)
  Interventions: Drug: Gefitinib

INTERVENTIONS:
Drug: Gefitinib — ZD1839 (gefitinib, IRESSA) 250 mg/DAY PO + 1 mg Anastrozole (ZD1033, Arimidex)
  Other Names: IRESSA
  Arms: Anastrozole-ZD1839
Drug: Anastrozole — 1 mg Anastrozole (ZD1033, Arimidex) + PLACEBO 1 TABLET/DAY PO
  Other Names: Arimidex
  Arms: Anastrozole-placebo

SUMMARY:
This study is being carried out to see if treatment with ZD1839 (Gefitinib) combined with Arimidex (Anastrozole) has improved efficacy over Arimidex alone in preventing progression of metastatic breast cancer.

DETAILED DESCRIPTION:
This is a phase II, multicenter, double-blind, randomized, placebo-controlled trial. Patients will be randomized in a double-blind manner in a 1:1 ratio to receive either 250 mg/day ZD1839 or matched placebo in combination with 1 mg/day anastrozole. The dose of ZD1839 has been selected based on clinical studies in other tumor types suggesting identical efficacy together with a better toxicity profile in patients treated at 250 mg compared to 500 mg/day. The 1 mg dose of anastrozole is the standard approved dose.

ELIGIBILITY:
Inclusion Criteria:

* Female postmenopausal patients aged 18 years or older with newly diagnosed metastatic breast cancer.
* Patients with recurrent disease during or after adjuvant tamoxifen or patients who are hormone therapy naïve are eligible for this trial.
* A paraffin embedded tumor tissue block or slides from either the metastatic or primary tumor site is required.

Exclusion Criteria:

* Patients cannot be on hormone replacement therapy while on study.
* Prior chemotherapy received for metastatic disease is not allowed.
* Previous treatment with tyrosine kinase inhibitors or aromatase inhibitors is not allowed.
* Patients who have evidence of an active interstitial lung disease are not eligible.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Estimated)
Dates: Start 2004-01; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Time to progression | Duration of study
  To estimate TTP in the 2 treatment arms of postmenopausal patients with newly diagnosed metastatic breast cancer

SECONDARY OUTCOMES:
Objective response rate | Duration of Study
  To estimate the ORR (complete response [CR] and partial response [PR] as defined by RECIST for the 2 treatment arms
Overall clinical benefit rate | Duration of Study
  To estimate the clinical benefit rates (CBR; defined as CR+PR[as per RECIST]+stable disease [SD]>24 weeks) for the 2 treatment arms
Overall survival | Duration of Study
  To estimate overall survival (OS) for each of the 2 treatment arms
Safety | Duration of Study
  To compare the tolerability of anastrozole/placebo to that of anastrozole/ZD1839
Pharmacokinetic variables | Duration of Study
  To determine steady-state plasma trough concentrations of anastrozole in all patients. To determine steady-state trough concentrations of ZD1839 and to relate values to historical data
Biomarker objectives | Duration of Study
  To obtain tumor tissue and blood samples for biologic studies in the limited population available and measure expression of markers that may potentially correlate with response to treatment in this patient population

CONTACTS AND LOCATIONS:
Overall Officials: Iressa Medical Science Director, MD, Study Director — AstraZeneca
Locations (27):
- United States (16):
  - Research Site, La Jolla, California
  - Research Site, San Diego, California
  - Research Site, Orlando, Florida
  - Research Site, Lafayette, Louisiana
  - Research Site, Rockville, Maryland
  - Research Site, Columbia, Missouri
  - Research Site, Omaha, Nebraska
  - Research Site, Las Vegas, Nevada
  - Research Site, Voorhees Township, New Jersey
  - Research Site, Albuquerque, New Mexico
  - Research Site, Lake Success, New York
  - Research Site, Cincinnati, Ohio
  - Research Site, Allentown, Pennsylvania
  - Research Site, Sioux Falls, South Dakota
  - Research Site, Houston, Texas
  - Research Site, Temple, Texas
- Research Site, Cali, Colombia
- Mexico (3):
  - Research Site, Aguascalientes
  - Research Site, Guadalajara
  - Research Site, Morelia
- Venezuela (7):
  - Research Site, Barcelona
  - Research Site, Barquisimeto
  - Research Site, Caracas
  - Research Site, Maracaibo
  - Research Site, Puerto Ordaz and San Felix
  - Research Site, San Cristóbal
  - Research Site, Valencia

REFERENCES:
- See also: CSR-1839US-0713.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=1553&filename=CSR-1839US-0713.pdf